CLINICAL TRIAL: NCT02247973
Title: PhaseⅡTrial of Co-transplantation With Bone Marrow Derived Mesenchymal Stem Cells From Related Donors in Alternative Donor Transplantation of Severe Aplastic Anemia.
Brief Title: Mesenchymal Stem Cells Co-transplantation in Alternative Donor Transplantation of Severe Aplastic Anemia.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Guangzhou General Hospital of Guangzhou Military Command (Other)
Collaborators: Guangzhou First People's Hospital (Other); Nanfang Hospital, Southern Medical University (Other); Southern Medical University, China (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Second Affiliated Hospital, Sun Yat-Sen University (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Fifth Affiliated Hospital, Sun Yat-Sen University (Other); Guangdong Provincial People's Hospital (Other); The Second People's Hospital of GuangDong Province (Other); First Affiliated Hospital of Jinan University (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); Second Affiliated Hospital of Guangzhou Medical University (Other); Peking University Shenzhen Hospital (Other); Shenzhen Second People's Hospital (Other)
Responsible Party: Principal Investigator, Yang Xiao, PhaseⅡtrial of co-transplantation with bone marrow derived mesenchymal stem cells from related donors in alternative donor transplantation of severe aplastic anemia., Guangzhou General Hospital of Guangzhou Military Command
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MSC-alternative donor SCT-SAA
Record Dates: First submitted 2014-09-17; First posted 2014-09-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Severe Aplastic Anemia
MeSH Terms: conditions — Anemia, Aplastic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mesenchymal stem cells (Experimental): Intravenous bone marrow derived mesenchymal stem cells infusion from related donor to patients with severe aplastic anemia.
  Interventions: Biological: mesenchymal stem cells

INTERVENTIONS:
Biological: mesenchymal stem cells — Intravenous administration of up to 1~2x10^6 MSCs per kg,for 2 times,d0 and d14
  Other Names: Multipotent Mesenchymal Stromal Cells
Biological: mesenchymal stem cells — bone marrow derived mesenchymal stem cells from related donors.

SUMMARY:
The study is a phase II trial designed to evaluate the efficacy and safety of co-transplantation with bone marrow derived mesenchymal stem cells from related donors in alternative donor transplantation of severe aplastic anemia.

DETAILED DESCRIPTION:
Aplastic anemia (AA) is an autoimmune hematologic stem cell disease mediated by activated T-lymphocytes that leads to bone marrow dysfunction. In the presence of an empty marrow, pancytopenia, and transfusion dependence, the severity of the disease is based on neutrophil (PMN) count: nonsevere AA (nSAA; PMN > 0.5 × 109/L), severe AA (SAA;PMN 0.2- 0.5 × 109/L), and very severe AA (vSAA; PMN< 0.2 × 109/L).

Allogeneic BMT from an HLA-identical sibling donor or matched-alternative donor is the treatment of choice for patients with aplastic anaemia.Transplantation for patients with severe aplastic anaemia from an HLA identical sibling donor is now very successful with a 75-90% chance of long term cure and with overall survival of between 65% and 73% at 5 years for matched-alternative donor transplantation. However, these two approachs are limited by the availability of HLA-matched donors.

Patients without HLA-identical sibling donor or matched-alternative donor can be offered immunosuppressive treatment (IST) involving injections of Anti-thymocyte globulin (ATG) in combination with cyclosporine (CsA). The treatment response with ATG is at best between 60-80%, 30%-40% patients relapse following an initial response to treatment. Moreover, a recent study has shown that on multivariate analysis of response at 6 months, only younger age, absolute reticulocyte count (ARC) and absolute lymphocyte count (ALC), correlate with response to ATG. Patients with SAA or vSAA, with much lower ARC and ALC, were poor response to IST and have high risks of dying of infection and bleeding.

Nowadays, with advances in transplant technology, HLA-mismatched related donors and unrelated donors transplantation has achieved good clinical results. Data from the XJ Huang indicated that patients with HLA-mismatched related donors achieved 100% donor myeloid engraftment and have a survival rate of 64.6±12.4%. Retrospectively analyzed results for 154 patients with acquired SAA who received BMT from unrelated donors identified through the Japan Marrow Donor Program showed the probability of OS at 5 years was 56% (95% confidence interval, 34%-78%).

Compared with malignant disease, mismatched related donor or unrelated donor HSCT for SAA involves distinct challenges mainly associated with high graft failure and high GVHD. So, if we can find a way to promote implantation meanwhile prevent or reduce GVHD , the efficacy of HLA-mismatched related donors transplantation can improve.

Mesenchymal stem cells (MSCs) are multi-potent non-hematopoietic progenitors mainly found in BM, cord blood, and adipose tissue. MSCs are attractive because of the ease with which they can be isolated and expanded ex vivo, their ability to undergo multilineage differentiation, and their lack of immunogenicity. These cells were shown to provide support for the growth and differentiation of hematopoietic progenitor cells in BM micro-environments. In additon, preliminary studies have shown clinical effectiveness of allogeneic MSC in the treatment of refractory graft-versus-host disease and an improvement in or resolution of severe aGVHD when co-transplantation with MSCs. Due to these properties, MSCs have become an interesting candidate for use in cellular therapy and are considered "theoretically perfect cells" for potential clinical use against AA mismatched related donors transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. In line with the 2009 Edition (United Kingdom) aplastic anemia diagnostic criteria for SAA or VSAA;
2. Age less than 50 years old,willing to transplant；
3. No HLA-identical sibling donor；
4. Have HLA-mismatched related donors or unrelated donors ( ≥5/10 HLA matched loci in related donors; ≥8/10 HLA matched loci in unrelated donors )
5. No serious infection or acute hemorrhage;
6. Cardiac ultrasound examination showed left ventricular ejection fraction is greater than 50%;
7. Both transaminase and serum creatinine level are no more than twice times the upper limit of normal value (ULN);
8. No acute infectious disease;
9. Ability to understand and the willingness to sign a written informed consent document.
10. ECOG score of 0-2 points.

Exclusion Criteria:

1. Patients with severe infection or active bleeding;
2. With severe cardiac insufficiency, left ventricular ejection fraction <50%;
3. With severe liver dysfunction, liver function (ALT and the TBIL) is higher than the ULN 3 times;
4. With severe renal insufficiency, renal function (Cr) is twice higher than the ULN; or 24-hour urine creatinine clearance rate (Ccr) lower than 50ml/min;
5. Active tuberculosis, severe acute hepatitis and other infectious diseases in active period;
6. ECOG score more than 3 points;
7. Accompanied by malignant tumors and other clonal disease;
8. Poor compliance and the researchers considered unsuitable for MSC infusion.

Ages: 14 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-02; Primary Completion 2017-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
survival rate | up to 2 years after HSCT
  The 2-year disease-free survival and overall survival.

SECONDARY OUTCOMES:
acute GVHD | UP to 3 months after HSCT
  The incidence of acute GVHD after HSCT.
chronic GVHD | UP to 2 years after HSCT
  The incidence of chronic GVHD after HSCT.
Transplant-related mortality | UP to 1 months after HSCT
Rates of relapse | UP to 2 years after HSCT
The implantation | Up to 4 weeks after HSCT
  The implantation rate and implantation time.

CONTACTS AND LOCATIONS:
Overall Officials: Yang Xiao, MD, Study Chair — Guangzhou General Hospital of Guangzhou Military Command
Locations (1):
- Guangzhou General Hospital of Guangzhou Military Command, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Marsh JC, Ball SE, Cavenagh J, Darbyshire P, Dokal I, Gordon-Smith EC, Keidan J, Laurie A, Martin A, Mercieca J, Killick SB, Stewart R, Yin JA; British Committee for Standards in Haematology. Guidelines for the diagnosis and management of aplastic anaemia. Br J Haematol. 2009 Oct;147(1):43-70. doi: 10.1111/j.1365-2141.2009.07842.x. Epub 2009 Aug 10. No abstract available. PMID 19673883
- [Background] Bacigalupo A, Locatelli F, Lanino E, Marsh J, Socie G, Maury S, Prete A, Locasciulli A, Cesaro S, Passweg J; Severe Aplastic Anemia Working Party of the European Group for Blood and Marrow Transplantation. Fludarabine, cyclophosphamide and anti-thymocyte globulin for alternative donor transplants in acquired severe aplastic anemia: a report from the EBMT-SAA Working Party. Bone Marrow Transplant. 2005 Dec;36(11):947-50. doi: 10.1038/sj.bmt.1705165. PMID 16205733
- [Background] Deeg HJ, O'Donnell M, Tolar J, Agarwal R, Harris RE, Feig SA, Territo MC, Collins RH, McSweeney PA, Copelan EA, Khan SP, Woolfrey A, Storer B. Optimization of conditioning for marrow transplantation from unrelated donors for patients with aplastic anemia after failure of immunosuppressive therapy. Blood. 2006 Sep 1;108(5):1485-91. doi: 10.1182/blood-2006-03-005041. Epub 2006 May 9. PMID 16684959
- [Background] George B, Mathews V, Viswabandya A, Lakshmi KM, Srivastava A, Chandy M. Allogeneic hematopoietic stem cell transplantation is superior to immunosuppressive therapy in Indian children with aplastic anemia--a single-center analysis of 100 patients. Pediatr Hematol Oncol. 2010 Mar;27(2):122-31. doi: 10.3109/08880010903540542. PMID 20201693
- [Background] Kojima S, Matsuyama T, Kato S, Kigasawa H, Kobayashi R, Kikuta A, Sakamaki H, Ikuta K, Tsuchida M, Hoshi Y, Morishima Y, Kodera Y. Outcome of 154 patients with severe aplastic anemia who received transplants from unrelated donors: the Japan Marrow Donor Program. Blood. 2002 Aug 1;100(3):799-803. doi: 10.1182/blood.v100.3.799. PMID 12130489
- [Background] Noort WA, Kruisselbrink AB, in't Anker PS, Kruger M, van Bezooijen RL, de Paus RA, Heemskerk MH, Lowik CW, Falkenburg JH, Willemze R, Fibbe WE. Mesenchymal stem cells promote engraftment of human umbilical cord blood-derived CD34(+) cells in NOD/SCID mice. Exp Hematol. 2002 Aug;30(8):870-8. doi: 10.1016/s0301-472x(02)00820-2. PMID 12160838
- [Background] Le Blanc K, Rasmusson I, Sundberg B, Gotherstrom C, Hassan M, Uzunel M, Ringden O. Treatment of severe acute graft-versus-host disease with third party haploidentical mesenchymal stem cells. Lancet. 2004 May 1;363(9419):1439-41. doi: 10.1016/S0140-6736(04)16104-7. PMID 15121408
- [Background] Ringden O, Uzunel M, Rasmusson I, Remberger M, Sundberg B, Lonnies H, Marschall HU, Dlugosz A, Szakos A, Hassan Z, Omazic B, Aschan J, Barkholt L, Le Blanc K. Mesenchymal stem cells for treatment of therapy-resistant graft-versus-host disease. Transplantation. 2006 May 27;81(10):1390-7. doi: 10.1097/01.tp.0000214462.63943.14. PMID 16732175
- [Background] Le Blanc K, Frassoni F, Ball L, Locatelli F, Roelofs H, Lewis I, Lanino E, Sundberg B, Bernardo ME, Remberger M, Dini G, Egeler RM, Bacigalupo A, Fibbe W, Ringden O; Developmental Committee of the European Group for Blood and Marrow Transplantation. Mesenchymal stem cells for treatment of steroid-resistant, severe, acute graft-versus-host disease: a phase II study. Lancet. 2008 May 10;371(9624):1579-86. doi: 10.1016/S0140-6736(08)60690-X. PMID 18468541
- [Background] Ball LM, Bernardo ME, Roelofs H, Lankester A, Cometa A, Egeler RM, Locatelli F, Fibbe WE. Cotransplantation of ex vivo expanded mesenchymal stem cells accelerates lymphocyte recovery and may reduce the risk of graft failure in haploidentical hematopoietic stem-cell transplantation. Blood. 2007 Oct 1;110(7):2764-7. doi: 10.1182/blood-2007-04-087056. Epub 2007 Jul 16. PMID 17638847
- [Background] Fang B, Li N, Song Y, Li J, Zhao RC, Ma Y. Cotransplantation of haploidentical mesenchymal stem cells to enhance engraftment of hematopoietic stem cells and to reduce the risk of graft failure in two children with severe aplastic anemia. Pediatr Transplant. 2009 Jun;13(4):499-502. doi: 10.1111/j.1399-3046.2008.01002.x. Epub 2008 Jul 30. PMID 18673358
- [Background] Wang H, Wang Z, Xue M, Liu J, Yan H, Guo Z. Co-transfusion of haplo-identical hematopoietic and mesenchymal stromal cells to treat a patient with severe aplastic. Cytotherapy. 2010 Jul;12(4):563-5. doi: 10.3109/14653241003695059. PMID 20380540
- [Background] Jaganathan BG, Tisato V, Vulliamy T, Dokal I, Marsh J, Dazzi F, Bonnet D. Effects of MSC co-injection on the reconstitution of aplastic anemia patient following hematopoietic stem cell transplantation. Leukemia. 2010 Oct;24(10):1791-5. doi: 10.1038/leu.2010.164. Epub 2010 Aug 19. No abstract available. PMID 20724985
- [Background] Fang B, Song Y, Li N, Li J, Han Q, Zhao RC. Mesenchymal stem cells for the treatment of refractory pure red cell aplasia after major ABO-incompatible hematopoietic stem cell transplantation. Ann Hematol. 2009 Mar;88(3):261-6. doi: 10.1007/s00277-008-0599-0. Epub 2008 Sep 4. PMID 18769919
- [Background] Xiao Y, Jiang ZJ, Pang Y, Li L, Gao Y, Xiao HW, Li YH, Zhang H, Liu Q. Efficacy and safety of mesenchymal stromal cell treatment from related donors for patients with refractory aplastic anemia. Cytotherapy. 2013 Jul;15(7):760-6. doi: 10.1016/j.jcyt.2013.03.007. PMID 23731760